CLINICAL TRIAL: NCT01082016
Title: Sleep Promotion in Critically Ill and Injured Patients Cared for in the Intensive Care Unit
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Arizona (Other)
Collaborators: Arizona Biomedical Research Commission (ABRC) (Other)
Responsible Party: Randall Friese, MD Associate Professor of Surgery, University of Arizona College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: ABRC 9-022
Record Dates: First submitted 2010-03-04; First posted 2010-03-05 (Estimated); Last update posted 2010-09-20 (Estimated); Status verified 2010-03

CONDITIONS: Sleep Deprivation
Keywords: Sleep; Critical Illness; Sleep promotion during recovery form illness
MeSH Terms: conditions — Sleep Deprivation; Critical Illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): Monitor sleep in ICU without attempts at promotion
- Sleep promotion (Experimental): Measure sleep in ICU with sleep promotion program in effect
  Interventions: Other: Sleep Enhancement Program (SEP)

INTERVENTIONS:
Other: Sleep Enhancement Program (SEP) — Sleep promotion in the ICU Multifaceted tool to promote sleep in ICU patients
  Arms: Sleep promotion

SUMMARY:
Sleep deprivation in healthy volunteers is associated with immune dysfunction. This adverse effect of sleep deprivation likely occurs in patients suffering from acute injury and critical illness requiring intensive care unit (ICU) admission. Studies have demonstrated that sleep in ICU patients is highly abnormal. The global hypothesis for this proposal is that a strategy to promote sleep in ICU patients will increase time in rapid eye movement (REM) and slow wave sleep (SWS). This three phase proposal examines the feasibility of a sleep promotion strategy for injured and critically ill patients in the ICU.

Phase I (Development and Training): Develop an intervention manual for sleep promotion, Sleep Enhancement Program (SEP), and train ICU staff.

Phase II (Validation and Safety): Implement SEP and test for protocol fidelity and safety.

Phase III (Efficacy): Conduct a pilot trail to determine efficacy of SEP to improve SWS in ICU patients.

ELIGIBILITY:
Inclusion Criteria:

* Received care in ICU for at least 3 days
* Received care in ICU no longer than 14 days
* Score of 3 to 5 on the Riker Sedation-Agitation Scale (SAS)
* Age < 55 years
* Able to tolerate PO or have gastric access present (Nasogastric/Orogastric/PEG)

Exclusion Criteria:

* Pregnancy
* Incarceration
* Admission diagnosis of Closed Head Injury or Traumatic Brain Injury
* Evidence of delirium on Confusion Assessment Method (CAM-ICU) Score
* Hemodynamic Instability
* Sepsis
* Multiple Organ Dysfunction
* Acute Renal Failure
* Known history of sleep disorder
* Known Psychiatric disorder

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Estimated)
Dates: Start 2010-04; Primary Completion 2013-01 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Time in Rapid Eye Movement (REM) Sleep | Within 24 hours of enrollment
  Polysomnography during sleep promotion protocol
Time in slow wave sleep | Within 24 hours of enrollment
  Polysomnography during sleep promotion protocol

SECONDARY OUTCOMES:
Systemic inflammatory mediators (cytokines) | Baseline and 12, 24, and 48 hours
  Blood draw for circulating mediaotors of inflammation
Safety profile | With 24 hours of enrollment
  Monitor for adverse events during polysomnography

CONTACTS AND LOCATIONS:
Overall Officials: Randall S Friese, MD, Principal Investigator — University of Arizona College of Medicine
Locations (1):
- University Medical Center, Tucson, Arizona, United States

REFERENCES:
- [Background] Parthasarathy S, Friese RS, Ayas NT. Biological validity to sleep measurements during critical illness. Crit Care Med. 2010 Feb;38(2):705-6. doi: 10.1097/CCM.0b013e3181cbb05f. No abstract available. PMID 20083935
- [Background] Friese RS. Good night, sleep tight: the time is ripe for critical care providers to wake up and focus on sleep. Crit Care. 2008;12(3):146. doi: 10.1186/cc6884. Epub 2008 May 12. PMID 18492219
- [Background] Friese RS, Diaz-Arrastia R, McBride D, Frankel H, Gentilello LM. Quantity and quality of sleep in the surgical intensive care unit: are our patients sleeping? J Trauma. 2007 Dec;63(6):1210-4. doi: 10.1097/TA.0b013e31815b83d7. PMID 18212640
- [Background] Friese RS. Sleep and recovery from critical illness and injury: a review of theory, current practice, and future directions. Crit Care Med. 2008 Mar;36(3):697-705. doi: 10.1097/CCM.0B013E3181643F29. PMID 18176314